# Comparison of Clinical Performance of Two Monthly Replacement Toric Soft Contact Lenses

**STUDY ID** 

CLV201-P003

**PROTOCOL** 

NCT06165627



#### **Device Protocol for CLV201-P003**

# Title: Comparison of Clinical Performance of Two Monthly Replacement Toric Soft Contact Lenses

Protocol Number: CLV201-P003

Clinical Investigation

Type:

Postmarket Interventional

Test Product: TOTAL30<sup>TM</sup> for Astigmatism (lehfilcon A)

Sponsor Name and Alcon Research, LLC, and its affiliates ("Alcon")

Address: 6201 South Freeway

Fort Worth, Texas 76134-2099

Property of Alcon Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Alcon

Document ID: V-CLN-0183501

\*\*

Status: Approved, Version: 3.0 Page 2 of 63 Approved Date: 15 Dec 2023

Investigator Agreement:

• I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices; applicable international and national regulations, laws, guidelines, and standards; the conditions of approval imposed by the reviewing IRB or regulatory authority; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.

- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current Investigator's brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical Investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authority? | | |
|---|---|---|---|
| | □ No | □Yes | |
| | Have you | ever been involved in a study or other research | that was terminated? |
| | □ No | □Yes | |
| | If yes, ple | ease explain here: | |
| Pr | incipal Inve | estigator: | |
| | | Signature | Date |
| | ame and prosition: | ofessional | |
| Αc | ddress: | | |

# **Table of Contents**

| De | evice Prote | ocol for CLV201-P003 | 1 |
|---|---|---|---|
| Ta | ble of Co | ntents | 3 |
| Li | st of Table | es | 5 |
| Li | st of Figu | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OI | F ACRONYMS AND ABBREVIATIONS | 13 |
| 3 | | COL SUMMARY | |
| 5 | INTROI | DUCTION | 26 |
| | 5.1 | Rationale and Background | 26 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | 27 |
| 6 | STUDY | OBJECTIVES | 28 |
| | 6.1 | Primary Objective(s) | 28 |
| | 6.2 | Secondary Objective(s) | 28 |
| | 6.3 | Safety Objective(s) | 28 |
| 7 | INVEST | TIGATIONAL PLAN | 28 |
| | 7.1 | Study Design | 28 |
| | 7.2 | Rationale for Study Design | 29 |
| | 7.3 | Rationale for Duration of Treatment/Follow-up | 29 |
| | 7.4 | Rationale for Choice of Comparator Product | 30 |
| 8 | STUDY | POPULATION | 30 |
| | 8.1 | Inclusion Criteria | 30 |
| | 8.2 | Exclusion Criteria | 31 |
| | 8.3 | Rescreening of Subjects | 33 |
| 9 | TREAT | MENTS ADMINISTERED | 33 |
| | 9.1 | Investigational Product(s) | 33 |
| | 9.2 | Other Medical Device or Medication Specified for Use During the Study | |
| | 9.3 | Treatment Assignment/Randomization | 36 |
| | 9.4 | Treatment Masking | 37 |

| | 9.5 | Accountability Procedures | 39 |
|---|---|---|---|
| | 9.6 | Changes to Concomitant Medications, Treatments/Procedures | 39 |
| 10 | STUDY | PROCEDURES AND ASSESSMENTS | 40 |
| | 10.1 | Informed Consent and Screening | 40 |
| | 10.2 | Description of Study Procedures and Assessments | |
| | | 10.2.1 Demographics | |
| | | 10.2.2 Medical History and Concomitant Medication | 41 |
| | | 10.2.3 Investigational Product Compliance | 41 |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 41 |
| | | 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment | 41 |
| | | 10.2.6 Device Deficiencies: Safety Assessment | 41 |
| | 10.3 | Unscheduled Visits | 42 |
| | 10.5 | Discontinued Subjects | 42 |
| | | 10.5.1 Screen Failures | 42 |
| | | 10.5.2 Discontinuations | 43 |
| | | 10.5.3 Schedule of Procedures and Assessments for Subjects | |
| | | Discontinued from Investigational Product | |
| | 10.6 | Clinical Study Termination. | 43 |
| | | 10.6.1 Follow-up of Subjects after Study Participation has Ended | |
| 11 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 44 |
| | 11.1 | General Information | 44 |
| | 11.2 | Monitoring for Adverse Events | 47 |
| | 11.3 | Procedures for Recording and Reporting | 47 |
| | 11.4 | Return Product Analysis | 49 |
| | 11.5 | Unmasking of the Study Treatment | 50 |
| | 11.6 | Follow-up of Subjects with Adverse Events | 50 |
| | 11.7 | | |
| 12 | ANALY | SIS PLAN | |
| | 12.1 | Subject Evaluability | 51 |
| | 12.2 | • | |
| | | 12.2.1 Safety Analysis Set | |
| | 12.3 | Demographic and Baseline Characteristics | |

| 12.4 | Effectiveness Analyses | 51 |
|-----------|----------------------------------------------------------|----|
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 52 |
| | 12.4.1.1 Statistical Hypotheses | 52 |
| | 12.4.1.2 Analysis Methods | 52 |
| 12.5 | Handling of Missing Data | 54 |
| 12.6 | Safety Analyses | 54 |
| 12.7 | Interim Analyses and Reporting | 55 |
| 13 DATA H | IANDLING AND ADMINISTRATIVE REQUIREMENTS | 55 |
| 13.1 | Subject Confidentiality | 55 |
| 13.2 | Completion of Source Documents and Case Report Forms | 55 |
| 13.3 | Data Review and Clarifications | 56 |
| 13.4 | Sponsor and Monitoring Responsibilities | 56 |
| 13.5 | Regulatory Documentation and Records Retention | 57 |
| 13.6 | Quality Assurance and Quality Control | 57 |
| 14 ETHICS | S | 58 |
| 15 REFERE | ENCES | 59 |
| 15.1 | Regulations and Standards | 59 |
| 15.2 | Scientific and Other References | 60 |
| | List of Tables | |
| Table 2–1 | List of Acronyms and Abbreviations Used in This Protocol | 13 |
| Table 3–1 | Schedule of Study Procedures and Assessments | 21 |
| Table 6–1 | Primary Objective(s) | 28 |
| Table 6–2 | Safety Objective(s) | 28 |
| Table 9–1 | Test Product | 33 |
| Table 9–2 | Comparator Product | 35 |

# **List of Figures**

| Figure 11-1 | Categorization of All Adverse Events | 45 |
|-------------|----------------------------------------------|----|
| Figure 11-2 | Categorization of All Serious Adverse Events | 45 |

# 1 GLOSSARY OF TERMS

| Names of Test Product(s) | Throughout this document, test product(s) will be referred to as TOTAL30 for Astigmatism (lehfilcon A) soft contact lenses |
|---|---|
| Name of Comparator<br>Product(s) | CooperVision® Biofinity® Toric (comfilcon A) soft contact lenses (No Biofinity Toric XR) |
| Adverse Device Effect (ADE) | Adverse event related to the use of an investigational medical device or comparator. |
| | Note: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation; any malfunction; and use error or intentional misuse. |
| Adverse Event (AE) | Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device or comparator and whether anticipated or unanticipated. |
| | Note: For subjects, this definition includes events related to the investigational medical device, comparator, or the procedures involved. For users or other persons, this definition is restricted to the use of the investigational medical device or comparator. |
| | Requirements for reporting adverse events in the study can be found in Section 11. |
| Anticipated Serious Adverse Device Effect (ASADE) | An effect which by its nature, incidence, severity, or outcome has been identified in the risk assessment. |
| Clinical Investigation Plan | The document(s) stating the rationale, objectives, design, |

| (CIP) | and prespecified analysis, methodology, organization, monitoring, conduct, and record-keeping of the clinical investigation. Note: The protocol and other documents referenced in the protocol (for example, the statistical analysis plan, the manual of procedures, the deviations and evaluability plan, and the protocol monitoring plan) comprise the CIP. |
|---|---|
| Clinical Investigation Report (CIR)/Clinical Study Report | The document describing the design, execution, statistical analysis, and results of a clinical investigation. The clinical investigation report is synonymous with the clinical study report. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance. Note: This definition includes malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling related to the investigational medical device or the comparator. Requirements for reporting device deficiencies in the study can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for participation in the study. |
| Point of Enrollment | The time at which, following recruitment and before any clinical investigation-related procedures are undertaken, a subject signs and dates the informed consent form. |
| Interventional Clinical Trial | A pre- or postmarket clinical investigation where the assignment of a subject to a particular medical device is decided in advance by a clinical investigation plan, or diagnostic or monitoring procedures requested in the CIP are in addition to those available as normal clinical practice and burden the subject. |

| Investigational Product | A preventative (vaccine), a therapeutic (drug or biologic), device, diagnostic, or palliative used as a test or comparator product in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the authorized form, or when used for an unauthorized indication, or when used to gain further information about the authorized form. |
|---|---|
| Malfunction | Failure of an investigational medical device to perform in accordance with its intended purpose when used in accordance with the instructions for use or clinical investigation plan (CIP), or investigator's brochure (IB). |
| Noninterventional Study | Clinical investigation that draws inferences about the possible effect of an intervention on subjects, but the investigator has not assigned subjects into intervention groups based on a protocol and has not made any attempts to collect data on variables beyond those available throughout the course of normal clinical practice and burden to the subject. NOTE: The term "noninterventional" is synonymous with "observational." |
| Nonserious Adverse Event | Adverse event that does not meet the criteria for a serious adverse event. |
| Postmarketing / Postauthorization study | Any study conducted within the conditions laid down in product labelling and other conditions laid down for the marketing of the product or under normal conditions of use. A postmarketing study falls either within the definitions of an interventional or a noninterventional study and may also fall within the definition of a postapproval study. |
| Product Complaint | Any oral, electronic, or written communication that alleges deficiencies related to the identity (labeling), quality, durability, reliability, safety, effectiveness, or performance of a marketed product, including failure of the product, |

| Randomized Subject | labeling, or packaging to meet specifications, whether or not the product is related to or caused the alleged deficiency. A complaint may allege that an adverse event or medical device malfunction has occurred. |
|---|---|
| Kandonnized Subject | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |
| Serious Adverse Event (SAE) | Adverse event that led to any of the following: |
| (SILE) | • Death. |
| | • A serious deterioration in the health of the subject, users or other persons as defined by one or more of the following: |
| | a) a life-threatening illness or injury Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, i.e., it does not include an event which hypothetically might have caused death had it occurred in a more severe form. |
| | b) any potentially sight-threatening event or permanent impairment to a body structure or a body function including chronic diseases. |
| | <ul> <li>c) inpatient hospitalization or prolonged<br/>hospitalization.</li> </ul> |
| | d) a medical or surgical intervention to prevent a) or b). |
| | e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use. |
| | Fetal distress, fetal death, congenital abnormality or |

| | birth defect including physical or mental impairment. |
|---|---|
| | Note: Planned hospitalization for a preexisting condition, or<br>a procedure required by the CIP, without serious<br>deterioration in health, is not considered a serious adverse<br>event. |
| | Refer to Section 11 for additional SAEs. |
| Serious Health Threat | Signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users, or other persons, and that requires prompt remedial action for other subjects, users, or other persons. |
| | Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals. |
| Study Start | The start of the study is considered to coincide with the enrollment of the first patient. |
| Study Completion | The completion of the study is considered to coincide with the study-level last subject last visit or the decision to terminate the trial, whichever is later. |
| Unanticipated Serious Adverse Device Effect (USADE) | Serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the risk assessment. |
| Use Error | User action or lack of user action while using the medical device that leads to a different result than that intended by the manufacturer or expected by the user. Note: |
| | <ul><li>a) Use error includes the inability of the user to complete a task.</li><li>b) Use errors can result from a mismatch between the</li></ul> |

| Document ID: |
|---------------|
| V-CLN-0183501 |

Status: Approved, Version: 3.0 Page 12 of 63 Approved Date: 15 Dec 2023

| Vulnerable Subject | characteristics of the user, user interface, task, or use environment. c) Users might be aware or unaware that a use error has occurred. d) An unexpected physiological response of the patient is not by itself considered a use error. e) A malfunction of a medical device that causes an unexpected result is not considered a use error." An individual who is unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response. |
|---|---|
|---|---|

2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2–1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| ASADE | Anticipated serious adverse device effect |
| BCVA | Best corrected visual acuity |
| Biofinity Toric | CooperVision Biofinity Toric (comfilcon A) soft contact lenses (No |
| , | Biofinity Toric XR) |
| BVL | Blue-violet light |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CIP | Clinical investigation plan |
| CIR | Clinical investigation report |
| CL | Confidence limit |
| COL | Clinical Operations Lead |
| CRF | Case report form |
| CSM | Clinical Site Manager |
| CTT | Clinical Trail Team |
| D | Diopter |
| DEP | Data evaluability plan |
| DFU | Directions for use |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| EN | European Standard |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| IRT | Interactive Response Technology |
| ISO | International Organization for Standardization |
| LogMAR | Logarithm of the minimum angle of resolution |
| mm | millimeter |
| MOP | Manual of procedures |
| N/A | Not applicable |
| OD | Right eye |
| OS | Left eye |
| ~ | |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SLE | Slit lamp examination |
| SOP | Standard operating procedure |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------------|
| T30fA | TOTAL30 for Astigmatism (lehfilcon A) soft contact lenses |
| USA | United States of America |
| USADE | Unanticipated serious adverse device effect |
| UV | Ultraviolet |
| VA | Visual acuity |

# **3 PROTOCOL SUMMARY**

| Investigational | Device |
|---|---|
| product type | |
| ~ - | |
| Study type | Interventional |
| Investigational | Test Product: TOTAL30 for Astigmatism soft contact lenses |
| products | (T30fA; lehfilcon A) |
| | Comparator Product: CooperVision Biofinity Toric soft contact lenses (Biofinity Toric; comfilcon A) (No Biofinity Toric XR) |
| Purpose and Scientific | Purpose of the study: |
| Rationale for the | The purpose of this study is to assess the clinical performance of |
| Study | TOTAL30 for Astigmatism (T30fA) soft contact lenses with |
| | Biofinity Toric soft contact lenses |
| Brief Summary of the | The objective of this study is to evaluate the clinical |
| Protocol | performance of 2 toric lenses: T30fA and Biofinity Toric soft |
| | contact lenses in a 30-day trial |
| | . This will be a randomized (participants |
| | are placed into groups by chance) |
| | bilateral |
| | crossover (participants will wear both study lenses that are |
| | intended for astigmatism), double-masked (both participants and |
| | investigators do not know which study lens they are receiving), |
| | multicenter study. |
| | This study will include volunteer participants 18-45 years old |
| | who currently wear toric contact lenses (participants who |
| | already wear Biofinity Toric or Alcon brand toric soft contact |
| | lenses, or those who wear daily disposable contact lenses will be |
| | excluded from this study). The participants need to have worn |
| | their toric contact lenses for at least 5 days per week and at least |
| | 12 hours a day during the past 3 months to qualify for this study. |

| Objective(s) | The primary objective is to evaluate the clinical performance of TOTAL30 for Astigmatism (T30fA) soft contact lenses as compared to Biofinity Toric soft contact lenses. |
|---|---|
| | The safety objective is to describe the safety profile of the study products. |
| Endpoint(s) | Primary Effectiveness • Distance VA (logMAR; OD, OS) with study lenses at Day 30 |



Distance VA (logMAR) with habitual lenses Manifest refraction BCVA (logMAR distance with manifest refraction) Medical history/concomitant medication Safety **AEs** Biomicroscopy Device deficiencies **Study Design** This will be a prospective, randomized , bilateral, crossover, double-masked, multicenter study. Subjects will be expected to attend 5 office visits including screening. The total duration of the subject's participation in the study will be approximately 74 days. Subject is expected to wear each of the assigned study lenses (test and comparator lenses) for 30 days of bilateral wear (total of 60 days of lens wear). **Subject population** Volunteer subjects aged 18-45 years of age. Current habitual toric soft contact lens wearers, with at least 3 months of contact lens wearing experience (excluding any Biofinity Toric soft habitual contact lens wearers, Alcon Toric contact lens wearers, and habitual daily disposable lens wearers). Wear habitual lenses at least 5 days per week and at least 12 hours per day during the past 3 months. To qualify, subjects must be able to wear contact lenses within a range of sphere & cylinder power and axes (Sphere:

Status: Approved, Version: 3.0

Approved Date: 15 Dec 2023

| | -0.50 D to -6.00 D in 0.25 D steps; Cylinder: -0.75 D and -1.25 D; Axis: 10°, 80°, 90°, 100°, 170°, 180°). Planned number of subjects enrolled/consented: ~ 66 Planned number of completed subjects: 60 |
|---|---|
| Sites and Locations | Planned number of clinical sites: ~ 5 Planned locations (initial list of locations, which may change during start up or conduct according to study needs): United States |
| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Successful wearer of toric soft contact lenses in both eyes for a minimum of 5 days per week and at least 12 hours per day during the past 3 months.</li> <li>Best corrected distance visual acuity (as determined by manifest refraction at screening) better than or equal to 0.10 logMAR in each eye.</li> <li>Able to wear contact lenses within a range of sphere &amp; cylinder power and axes (Sphere: -0.50 D to -6.00 D in 0.25 D steps; Cylinder: -0.75 D and -1.25 D; Axis: 10°, 80°, 90°, 100°, 170°, 180°).</li> </ul> |
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) | <ul> <li>Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates.</li> <li>Monovision and multifocal contact lens wearers.</li> <li>Habitual Biofinity Toric soft contact lens wearers, daily disposable contact lens wearers, and Alcon Toric contact lens wearers in the past 3 months prior to consent.</li> <li>Wearing habitual contact lenses in extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment</li> </ul> |



Table 3-1 Schedule of Study Procedures and Assessments

| | | LENS 1<br>(Period 1) | | LENS 2<br>(Period 2 | | | |
|---|---|---|---|---|---|---|---|
| | Visit 1<br>Screen/Baseline/<br>Lens Fitting | Visit 2<br>Dispense Lens 1 | Visit 3<br>Day 30<br>Follow-<br>up Lens<br>1 | Visit 4 Dispense<br>Lens 2 | Visit 5<br>Day 30<br>Follow-up<br>Lens<br>2/Exit | Unscheduled<br>visit | Early<br>Exit |
| Procedure/Assessment | | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 1] | Day 30<br>(-1/+3)<br>Days | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 3] | Day 30<br>(-1/+3)<br>Days | N/A | N/A |
| Informed Consent | X | | | | | | |
| Demographics | X | | | | | | |
| Medical History | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X |
| Habitual lens information (brand, lens power*, lens care*) | X | | | | | | |
| VA with habitual correction<br>(spectacles or contact lenses) (OD,<br>OS, Snellen distance)* | X | | | | X | (X) | X |
| Keratometry (OD, OS) * | X | | | | | | |
| Manifest refraction* | X | (X) | (X) | (X) | (X) | (X) | (X) |

| | | LENS 1<br>(Period 1) | | LENS 2<br>(Period 2 | | | |
|---|---|---|---|---|---|---|---|
| | Visit 1<br>Screen/Baseline/<br>Lens Fitting | Visit 2<br>Dispense Lens 1 | Visit 3<br>Day 30<br>Follow-<br>up Lens<br>1 | Visit 4 Dispense<br>Lens 2 | Visit 5<br>Day 30<br>Follow-up<br>Lens<br>2/Exit | Unscheduled<br>visit | Early<br>Exit |
| Procedure/Assessment | | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 1] | Day 30<br>(-1/+3)<br>Days | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 3] | Day 30<br>(-1/+3)<br>Days | N/A | N/A |
| BCVA* (OD, OS, logMAR distance with manifest refraction) | X | (X) | (X) | (X) | (X) | (X) | (X) |
| Biomicroscopy | X | X | X | X | X | X | X |
| Inclusion/Exclusion | X | | | | | | |
| Lens Fitting (Test and Comparator)<br>fitting and evaluation* (logMAR<br>VA and lens fitting assessments) | X | | | | | | |
| Determine study lens power parameters* | X | | | | | | |
| Randomization | X | | | | | | |
| Determine final study lens power parameters to be dispensed | | X | | X | | | |

LENS 2

Status: Approved, Version: 3.0 Approved Date: 15 Dec 2023

LENS 1

| | | (Period 1) | | (Period 2) | | | | |
|---|---|---|---|---|---|---|---|---|
| | Visit 1<br>Screen/Baseline/<br>Lens Fitting | Visit 2<br>Dispense Lens 1 | Visit 3<br>Day 30<br>Follow-<br>up Lens<br>1 | Visit 4 Dispense<br>Lens 2 | Visit 5<br>Day 30<br>Follow-up<br>Lens<br>2/Exit | Unscheduled<br>visit | Early<br>Exit | |
| Procedure/Assessment | | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 1] | Day 30<br>(-1/+3)<br>Days | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 3] | Day 30<br>(-1/+3)<br>Days | N/A | N/A | |
| Dispense study lenses* | | X | | X | | | | 1 |
| VA w/study lenses (OD, OS, logMAR distance) | | x | X | х | X | (X) | (X) | |

| | | LENS 1<br>(Period 1) | | LENS 2<br>(Period 2 | | | |
|---|---|---|---|---|---|---|---|
| | Visit 1<br>Screen/Baseline/<br>Lens Fitting | Visit 2<br>Dispense Lens 1 | Visit 3<br>Day 30<br>Follow-<br>up Lens<br>1 | Visit 4 Dispense<br>Lens 2 | Visit 5<br>Day 30<br>Follow-up<br>Lens<br>2/Exit | Unscheduled<br>visit | Early<br>Exit |
| Procedure/Assessment | | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 1] | Day 30<br>(-1/+3)<br>Days | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 3] | Day 30<br>(-1/+3)<br>Days | N/A | N/A |
| Lens Wear Calendar * | | Dispense | Collect | Dispense | Collect | | Collect |
| Collect Worn Lenses * | | | X | | X | (X) | X |

| | | LENS 1<br>(Period 1) | | LENS 2<br>(Period 2) | | | |
|---|---|---|---|---|---|---|---|
| | Visit 1<br>Screen/Baseline/<br>Lens Fitting | Visit 2<br>Dispense Lens 1 | Visit 3<br>Day 30<br>Follow-<br>up Lens<br>1 | Visit 4 Dispense<br>Lens 2 | Visit 5<br>Day 30<br>Follow-up<br>Lens<br>2/Exit | Unscheduled<br>visit | Early<br>Exit |
| Procedure/Assessment | | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 1] | Day 30<br>(-1/+3)<br>Days | Day 1 [2 Days (at least 48 hours)-4 Days Washout period with habitual spectacles only after Visit 3] | Day 30<br>(-1/+3)<br>Days | N/A | N/A |
| Adverse Events | X | X | X | X | X | X | X |
| Device deficiencies | X | X | X | X | X | X | X |
| Exit Form | (X) | (X) | (X) | (X) | X | | X |

<sup>(</sup>X) assessment performed as necessary, e.g., decrease of VA by 2 lines or more with investigational product (IP)

<sup>\*</sup> Source only and transferred to the sponsor upon request



#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the study sponsor and must be approved by the IRB/IEC and global and regional health authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### **5 INTRODUCTION**

# 5.1 Rationale and Background

T30fA are a new monthly replacement soft contact lenses, which utilize water gradient technology, and contain 55% water content at the core that gradually increases to nearly 100% at the outer surface. The lenses also use biomimetic Celligent Technology, which has properties that allow the lens to mimic the corneal surface. The innovative surface chemistry provides an extremely soft and lubricious lens surface and helps to resist bacterial and lipid deposit adhesion. T30fA contact lenses also offer UV and blue-violet light (BVL) filtering. T30fA lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia, with astigmatism) in persons with nondiseased eyes.

#### **5.2** Purpose of the Study

The purpose of this study is to assess the clinical performance of T30fA contact lenses compared to the commercially available Biofinity Toric soft contact lenses

The endpoints have been selected to address the primary objective of the study. Procedures for measurement of these endpoints were selected based on common practice for these assessments. The design of this study is justified based upon preclinical and clinical testing, as described within the package insert. Biofinity Toric soft contact lenses were chosen as the comparator product because these lenses have the same wear modality and replacement schedule.

The lenses are intended for daily wear (less than 24 hours while awake), with removal for cleaning and disinfection (chemical, not heat) prior to reinsertion, or disposal, as recommended by the eye care professional. Lenses should be discarded and replaced after one month.

There are no immediate plans to submit the results of this study for publication; however, the results may be offered for publication if they are of scientific interest, or if the results relate to a product that is subsequently approved or cleared for marketing.

#### 5.3 Risks and Benefits

The clinical investigation process risks are managed through appropriate training and monitoring according to the protocol-specific monitoring plan. Investigational device risks, including risks associated with use of device and methods and procedures for application of device, are defined in the investigator's brochure and/or product labeling and are managed through review of safety assessments outlined in this protocol.

T30fA (lehfilcon A) soft contact lenses and Biofinity Toric contact lenses are commercially available for daily wear use under a frequent replacement wear modality; further details on any known potential risks and benefits can be found in the DFU.

A summary of the known potential risks and benefits associated with the T30fAand Biofinity Toric soft contact lenses can be found in the package insert. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, as well as through close clinical supervision by a licensed clinician during

exposure to the study lenses. The site personnel will educate subjects on proper hygiene and lens handling, as well as compliance with the use of contact lenses according to the protocol.

Refer to the package insert for additional information on risks and benefits.

#### 6 STUDY OBJECTIVES

#### 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| The objective of this study is to evaluate the clinical performance of TOTAL30 for Astigmatism (T30fA) soft contact lenses as compared to Biofinity Toric soft contact lenses | Distance VA (logMAR; OD, OS) with<br>study lenses at Day 30 |

#### 6.2 Secondary Objective(s)

Not applicable.

# 6.3 Safety Objective(s)

Table 6–2 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Describe the safety profile of the study products | <ul><li>Adverse events</li><li>Biomicroscopy findings</li><li>Device deficiencies</li></ul> |

#### 7 INVESTIGATIONAL PLAN

# 7.1 Study Design

This is a prospective, randomized, bilateral crossover, controlled, double-masked, clinical study to be conducted at approximately 5 sites. Eligible habitual toric soft contact lens wearers will be randomized to 1 of the 2 crossover sequences. Investigator and subject will be masked. A designated unmasked study staff member will prepare the contact lenses for dispensing.

Subjects will be expected to attend 5 office visits and will be dispensed study lenses (per randomization sequence) for 30-day duration of bilateral wear with each study lens (~60 days of lens wear).

the subject will wear the lenses each day for at least 12 hours per day.

At Visit 1 screening/baseline, lens fitting and randomization will be performed. Subject will return to the office for Visit 2 and Visit 4 after washout period (2-4 days) and will be dispensed their assigned study lens by an unmasked study staff member.

At Visit 3 and Visit 5 (Day 30 -1/+3 days) in-office lens fitting assessments for study lenses will be performed; once Visit 5 is complete subjects will exit from the study.



# 7.2 Rationale for Study Design

The crossover design will ensure that the same subject is exposed to both the test and comparator lens materials; therefore, objective assessments will be obtained for both lenses from the same subject. The study will include only those subjects who are current wearers of toric soft contact lenses in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week, and at least 12 hours per day. This will avoid confounding safety responses in nonadapted subjects. Furthermore, the subjects will not be permitted to use lubrication/rewetting drops during the duration of the study

# 7.3 Rationale for Duration of Treatment/Follow-up

The duration of product use is in accordance with product labeling.

#### 7.4 Rationale for Choice of Comparator Product

The Biofinity Toric soft contact lens was chosen as the comparator product as these lenses have the same wear modality and replacement schedule as T30fA.

#### **8 STUDY POPULATION**



#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

- 1. Subject must be 18-45 years old and must be able to understand and sign an IRB/IEC approved informed consent form.
- 2. Willing and able to attend all scheduled study visits as required per protocol.
- 3. Successful wearer of toric soft contact lenses in both eyes for a minimum of 5 days per week and at least 12 hours per day during the past 3 months.
- 4. Best corrected distance visual acuity (as determined by manifest refraction at screening) better than or equal to 0.10 logMAR in each eye.
- 5. Able to wear contact lenses within a range of sphere and cylinder power and axes (Sphere: -0.50 D to -6.00 D in 0.25 D steps; Cylinder: -0.75 D and -1.25 D; Axis: 10°, 80°, 90°, 100°, 170°, 180°).
- 6. Subject must be willing to stop wearing their habitual contact lenses for the duration of study participation.
- 8. Subject must possess spectacles and willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.
- 9. Subject must be willing to NOT use rewetting/lubricating drops and topical ocular medication at any time during study.

#### 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.

- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.
- 3. History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye.
- 4. Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study.
- 5. Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates.
- 6. Current or history of pathologically dry eye in either eye that, in the opinion of the investigator, would preclude contact lens wear.
- 7. Current or history of herpetic keratitis in either eye.
- 8. Eye injury in either eye within 12 weeks immediately prior to enrollment for this trial.
- 9. Current or history of intolerance, hypersensitivity or allergy to any component of the study products.
- 10. The investigator, his/her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of the aforementioned persons may not participate in the study.
- 11. Participation of the subject in a clinical trial within the previous 30 days or currently enrolled in any clinical trial.
- 12. Monovision and multifocal contact lens wearers.
- 13. Habitual Biofinity Toric/Biofinity Toric XR, daily disposable contact lens wearers, and Alcon Toric contact lens wearers in the past 3 months prior to consent.
- 14. Wearing habitual contact lenses in extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment
- 15. Currently pregnant, as stated by subject.

# 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

#### 9 TREATMENTS ADMINISTERED

# 9.1 Investigational Product(s)

Test Product(s): TOTAL30 for Astigmatism (lehfilcon A)

Comparator Product(s) (If applicable):

CooperVision Biofinity Toric (comfilcon A)

Table 9–1 Test Product

| TOTAL30 for Astigmatism (lehfilcon A) soft contact lenses |
|----------------------------------------------------------------------|
| Alcon Laboratories, Inc. |
| 6201 South Freeway |
| Fort Worth, Texas 76134-2099 |
| USA |
| TOTAL30 for Astigmatism (lehfilcon A) soft contact lenses are |
| indicated for the optical correction of ametropia (myopia or |
| hyperopia, with astigmatism) in persons with nondiseased eyes. |
| The lenses are intended for daily wear (less than 24 hours while |
| awake), with removal for cleaning and disinfection (chemical, not |
| heat) prior to reinsertion, or disposal, as recommended by the eye |
| care professional. Lenses should be discarded and replaced after one |
| month. |
| Material: lehfilcon A |
| Water content: 55% by weight in normal saline |
| Power range: |
| o Sphere: -0.50 to -6.00 D in 0.25 D steps |
| o Cylinder: -0.75 and -1.25 D |
| o Axis: 10°, 80°, 90°, 100°, 170°, 180° |
| Base curve (mm): 8.6 |
| • Diameter (mm): 14.5 |

| Formulation | Refer to the package insert/DFU for the lens material and package saline formulation. |
|---|---|
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> </ul> </li> <li>Replacement period: 30-day replacement</li> <li>Exposure: Subject duration of exposure to test lenses will be approximately 30 days and at least 12 hours per day.</li> <li>Lens Care: CLEAR CARE Cleaning &amp; Disinfecting Solution will be used during the duration of the study.</li> </ul> |
| Number/Amount of product to be provided to the subject | Each site will procure their own test lenses. |
| Packaging description | Provided in commercial packaging |
| Labeling description | Commercial foil |
| Training and/or experience requirements for device | No additional training or experience is required to administer the test product. |
| Storage conditions | Lenses are to be stored at room temperature. |
| Additional information | N/A |

| Supply | Site will procure the lenses which are commercially available. Refer |
|---|---|
| | to the MOP for a detailed description. |

Table 9–2 Comparator Product

| Comparator | Biofinity® Toric (comfilcon A) soft contact lenses |
|---|---|
| Product(s) | (No Biofinity Toric XR) |
| Manufacturer | CooperVision |
| Indication for Use | The intended use of this product is for vision correction. |
| Product description<br>and parameters<br>available for this<br>study | <ul> <li>Material: comfilcon A</li> <li>Water content: 48%</li> <li>Power range: <ul> <li>Sphere: -0.50 to -6.00 D in 0.25 D steps</li> <li>Cylinder: -0.75 and -1.25 D</li> </ul> </li> </ul> |
| | <ul> <li>Axis: 10°, 80°, 90°, 100°, 170°, 180°</li> <li>Base curve (mm): 8.7</li> <li>Diameter (mm):14.5</li> </ul> |
| Formulation | Refer to the package insert/DFU for the lens material and package saline formulation. |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> </ul> </li> <li>Replacement period: 30-day replacement</li> <li>Exposure: Subject duration of exposure to comparator lenses will be approximately 30 days and at least 12 hours per day.</li> <li>Lens Care: CLEAR CARE Cleaning &amp; Disinfecting Solution will be used during the duration of the study.</li> </ul> |
| Number/Amount of | Each site will procure their own comparator lenses. |
|---|---|
| Product to be | |
| Provided to the | |
| subject | |
| Packaging | Provided in commercial packaging |
| description | |
| Labeling description | Commercial foil |
| Training and/or | No additional training or experience is required to administer the |
| experience | test product. |
| requirements for | |
| device | |
| Storage conditions | Lenses are to be stored at room temperature. |
| Additional | N/A |
| identifying | |
| information | |
| Supply | Site will procure the lenses which are available commercially. Refer |
| | to the MOP for a detailed description. |

# 9.2 Other Medical Device or Medication Specified for Use During the Study

No other medical devices or medications are required to be used in conjunction with the treatments during the clinical study.

# 9.3 Treatment Assignment/Randomization

Qualified subjects will be randomized in a 1:1 ratio to receive treatment (lens) in crossover sequence: test product then comparator product or comparator product then test product, respectively.

Sequence 1: T30fA/Biofinity Toric

Sequence 2: Biofinity Toric/T30fA

Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

Status: Approved, Version: 3.0

Approved Date: 15 Dec 2023

A randomization list will be generated using a validated system that automates the random assignment of treatment arms to randomization numbers in the specified ratio. Subjects will be assigned treatment according to the randomization list uploaded in the randomization system. The randomization list will be generated and maintained by the study sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/randomization integration system to one of the treatments (lens sequences). The unmasked delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject randomization list but will not be communicated to the site user. The EDC/randomization integration system will inform the site user of the treatment (lens sequence) assignment to be dispensed to the subject.

## 9.4 Treatment Masking

This study is double-masked with subjects randomized in a 1:1 crossover manner for 30 days bilateral wear of T30fA soft contact lens and Biofinity Toric soft contact lens (total of 60 days of lens wear).





This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.



In the event of a medical emergency where the knowledge of subject treatment is required, an individual investigator will have the ability to unmask the treatment assignment for a specific subject after contacting an appropriate study sponsor representative if time allows.

Unmasking must be done according to the instructions provided for the study IRT system.

## 9.5 Accountability Procedures

Upon receipt of the IPs, the unmasked delegate must conduct an inventory, as applicable. During the study, designated unmasked study staff will provide the study lens to the subjects in accordance with their randomization assignment. Throughout the study, the unmasked delegate must maintain records of IP dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the investigator must be accounted for by study sponsor personnel, and in no case be used in an unauthorized situation.

The unmasked delegate should make every effort to collect used lenses and supplies from subjects.

It is the investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All unused products are available for return to the study sponsor, as directed
- Any study lenses, solutions associated with a device deficiency or with any productrelated adverse event (i.e., ADE or SADE) are returned to the study sponsor for
  investigation, unless otherwise directed by the sponsor. Refer to Section 11 of this
  protocol for additional information on the reporting of device deficiencies and AEs and
  the return of study products associated with these events.

The investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.

# 9.6 Changes to Concomitant Medications, Treatments/Procedures

After the subject is enrolled into the study, the investigator or site staff must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications
- Any medical procedure or hospitalization that occurred or is planned
- Any nondrug therapies (including physical therapy and blood transfusions)

The investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 5 office visits, as shown below.

| Visit # | Visit Type | Visit Window |
|---|---|---|
| Visit 1 | Screen/Baseline/Lens Fitting | N/A |
| Visit 2 | Dispense Lens 1 | 2 days (at least 48 hours) - 4 days<br>washout period with habitual spectacles<br>only after Visit 1 |
| Visit 3 | Day 30 Follow-up Lens 1 | Day 30 (-1/+3 days) |
| Visit 4 | Dispense Lens 2 | 2 days (at least 48 hours) - 4 days<br>washout period with habitual spectacles<br>only after Visit 3 |
| Visit 5 | Day 30 Follow-up Lens 2/Exit | Day 30 (-1/+3 days) |

Unscheduled visits and early exit visits are allowed, if necessary.

## 10.1 Informed Consent and Screening

The investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.

# 10.2 Description of Study Procedures and Assessments

Study-specific procedures and assessments described here may include standard of care; other standard of care procedures performed in the clinical management of the subject are not excluded.

Detailed descriptions of assessments and procedures are provided in the MOP. The investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

## 10.2.1 Demographics

Document ID:

Obtain demographic information including age, race, ethnicity, and sex.

## 10.2.2 Medical History and Concomitant Medication

Collect medical history information (within 1 year prior to screening visit), including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

Targeted Medical history and concomitant medications will be collected in the eCRF as outlined in the MOP.

## **10.2.3 Investigational Product Compliance**

Review subject compliance with the IP usage and adjunct product usage and collect all used and unused study IPs and other products that were dispensed.

## 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any adverse events that are observed or reported since the previous visit, including those associated with changes in concomitant medication dosing. See Section 11 for further details regarding AE collection and reporting.

# 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment

SLE of the cornea, iris/anterior chamber and lens must be performed in both eyes before instillation of any diagnostic eye drops.

# 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11. Note: AEs and device deficiencies must be recorded for all enrolled subjects from the time of signature of informed consent, regardless of subject enrollment status (screen failure or randomized).

#### **10.3** Unscheduled Visits

If a subject visit occurs between any regularly scheduled visit and the visit is conducted by study personnel, this visit must be documented as an Unscheduled Visit. If the subject seeks medical attention outside the clinic (for example, at an emergency room) or at the clinic but is seen by nonstudy personnel, the investigator is to capture adverse event-related information on the adverse event form upon becoming aware.

During all unscheduled visits, the investigator must conduct the following procedures:

- Collect adverse event information, as applicable
- Collect device deficiency information, as applicable
- Record changes in medical condition or concomitant medication
- Biomicroscopy

The investigator may perform additional procedures for proper diagnosis and treatment of the subject. The investigator must document this information in the subject's case history source documents.

If during an Unscheduled Visit the subject is discontinuing the IP or discontinuing from the study, the investigator must conduct Exit procedures according to Table 3–1 Schedule of Study Procedures and Assessments as possible.

# 10.4 Unplanned Lens Replacement

No spare lenses will be dispensed to the subject. If a lens is lost, damaged, or needs to be replaced due to a device deficiency/ADE, the subject will be instructed to return for an unplanned lens replacement. Refer to MOP for details.

# 10.5 Discontinued Subjects

#### 10.5.1 Screen Failures

Subjects who were excluded from the study after signing the informed consent and prior to randomization to product/dispense of study product.

The investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be reused.

#### 10.5.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the investigator after signing the informed consent.

Subject numbers of discontinued subjects must not be reused (i.e., subject replacement is not allowed).

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the investigator, continued treatment poses a risk to their health.

If a subject discontinues from study treatment, every effort must be made to keep the subject in the study and to continue with the study assessments as specified in the schedule of study procedures and assessments until the final visit.

For subjects discontinuing from the study, the investigator must complete all Exit procedures according to Table 3–1 Schedule of Study Procedures and Assessments and Section 10.5.3, if the subject is willing and able, and if in the opinion of the investigator it is safe for the subject to do so.

The investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.5.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an early exit visit. Refer to Table 3–1 and the MOP for details.

# 10.6 Clinical Study Termination

The study sponsor reserves the right to suspend or close the investigational site or suspend or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the study sponsor:

• The study sponsor must:

- o Immediately notify the investigator(s) and subsequently provide instructions for study termination.
- o Inform the investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for poststudy treatment options as needed.

The investigator may terminate the site's participation in the study for reasonable cause.

Breaking of the masked treatment codes will be done after locking the database.

## 10.6.1 Follow-up of Subjects after Study Participation has Ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11-1 Categorization of All Adverse Events



Figure 11-2 Categorization of All Serious Adverse Events



#### Serious Adverse Events

In addition to reporting all adverse events (serious and nonserious) meeting the definitions, the investigator must report any occurrence of the following as an SAE:

- An ocular infection, including a presumed infectious ulcer with any of the following characteristics:
  - Central or paracentral location
  - o Penetration of Bowman's membrane

- Infiltrates > 2 mm diameter
- o Iritis
- o Increase in intraocular pressure
- o Culture positive for microorganisms
- o Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon
- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from Baseline Visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

NOTE: For cultured events, document available results in the narrative section(s) of the corresponding ADE-SAE eCRF.

#### Other Ocular Adverse Events

The investigator must also report any ocular AE that is nonserious, device-related, nonsight threatening, and warrants discontinuation of any Contact Lens wear for greater than or equal to 2 weeks. The following are examples of such AEs:

- Peripheral nonprogressive noninfectious ulcers
- All symptomatic corneal infiltrative events
- Corneal staining score moderate (dense coalescent staining up to 2 mm) or greater
- Temporary vision loss as defined by loss of 2 or more lines of BCVA from baseline visit that persists for 2 or more weeks
- Neovascularization with vessel penetration of 1 mm or greater

The above events are based on the categories provided in the International Organization for Standardization (ISO) 11980 and the US FDA Premarket Notification (510(k)) Guidance Document for Daily Wear Contact Lenses and Contact Lens Care.

#### **Device Deficiencies**

A device deficiency may or may not be associated with subject harm (i.e., ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The investigator should determine the applicable category for the identified or suspect device deficiency and report any subject harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (e.g., incorrect lens power/diameter/base curve/color)
- Lens cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (e.g., mislabeled product)
- Suspect product contamination

## 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the investigator should inquire about AEs by asking the standard questions shown below and report as applicable:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

In addition, changes in any protocol-specific parameters evaluated during the study are to be reviewed by the investigator. Any untoward (unfavorable and unintended) change in a protocol-specific parameter that is clinically relevant, in the opinion of the investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

# 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any preexisting medical conditions or signs/symptoms present in a subject prior to the start of the study (i.e., before informed

consent is signed) are not considered AEs in the study and should be recorded in the medical history section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

For each recorded event, the ADEs and SAEs documentation must include date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the investigator must document all device deficiencies reported or observed with test and comparator products on the device deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the study sponsor immediately as follows:

- All SAEs must be reported immediately (within 24 hours) of the investigator's or site's awareness.
- ADEs that do not meet seriousness criteria and device deficiencies must be reported within 10 calendar days of the investigator's or site's awareness.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from discharge summary, autopsy report, certificate of death, etc., if applicable, in narrative section of the adverse device effect (for related AEs) and *Serious Adverse Event* eCRF.

Note: Should the EDC system become nonoperational, the site must complete the appropriate paper serious adverse event and adverse device effect and/or device deficiency form.

Study sponsor representatives may be contacted for any protocol-related question and their contact information is provided in the manual of procedures that accompanies this protocol.

Further, depending upon the nature of the AE or device deficiency being reported, the study sponsor may request copies of applicable portions of the subject's medical records. The investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

#### **Intensity and Causality Assessments**

Where appropriate, the investigator must assess the intensity (severity) of the AE based on medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the investigator must assess the causality (related or not related to the medical device or study procedure). An assessment of causality will also be performed by study sponsor utilizing the same definitions, as shown below:

#### Causality

Related An AE classified as related may be either definitely related or possibly related

where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that

the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply

unlikely to be related (i.e., there are other more likely causes for the AE).

The study sponsor will assess the AEs and may upgrade the investigator's assessment of seriousness and/or causality. The study sponsor will notify the investigator of any AE that is upgraded from nonserious to serious or from unrelated to related.

# 11.4 Return Product Analysis

Study sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.

#### 11.5 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study. If the treatment code needs to be broken in the interest of subject safety, the investigator is encouraged to contact an appropriate study sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (i.e., medical emergency), the code may be broken prior to contact with the study sponsor. The study sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the study sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements.

## 11.6 Follow-up of Subjects with Adverse Events

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The investigator should provide the study sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (i.e., database lock).

All complaints received after this time period will be considered and processed as spontaneous (following the post market vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements.

The investigator should also report complaints on non-Alcon products (i.e., Biofinity Toric) directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

# 11.7 Pregnancy in the Clinical Study

Women who are pregnant (as stated by subject) at the time of study entry are excluded from participation. However, pregnancy should be included in the Pregnancy eCRF if a woman becomes pregnant (as stated by the subject) during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, SD, median, minimum, and maximum, as well as CIs or CLs where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

Any deviations to this analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

## 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens sequence) assignment and locking the database, based upon the data evaluability plan (DEP).

## 12.2 Analysis Sets

## 12.2.1 Safety Analysis Set

| Safety analyses will be conducted using the safety analysis set on a treatment | nt-emergent basis |
|---|---|
| As such, the safety analysis set will include all subjects/eyes exposed to any | study lenses |
| evaluated in this study. | |
| | any AE or device |
| deficiency occurring after informed consent and prior to the initial exposure | to the study |
| lenses (test or comparator) under evaluation in this clinical protocol will be | listed as |
| pretreatment. | |

For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

# 12.3 Demographic and Baseline Characteristics

Demographic information will be summarized by lens sequence and overall. Frequencies and percentages will be presented for categorical variables such as sex, age group, race (race subgroups), and ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.

# 12.4 Effectiveness Analyses



## 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective is to evaluate the clinical performance of T30fA soft contact lenses as compared to Biofinity Toric soft contact lenses.

The primary endpoint is distance VA with study lenses at Day 30, collected for each eye, in logMAR.

## 12.4.1.1 Statistical Hypotheses

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.

## 12.4.1.2 Analysis Methods

Descriptive statistics will be provided as number of observations, mean, SD, median, minimum, and maximum.





## 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for effectiveness analyses.

## 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of AEs as well as the other listed parameters.

All AEs occurring from the time a subject signs the informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (frequencies and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation and SAEs will be identified. Individual subject listings will be provided, as necessary. Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Each biomicroscopy parameter will be tabulated by its grade. For each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (last assessment prior to study lens exposure) to any subsequent visit will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits for those eyes experiencing the increase.

Two listings for device deficiencies, prior to exposure to study lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be conducted for the safety analyses.

## 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

#### 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

## 13.1 Subject Confidentiality

The investigator must ensure that the subject's identity is kept confidential throughout the course of the study. In particular, the investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. The study sponsor may collect a copy of the enrollment log without any directly identifying subject information.

The study sponsor may share patient-level data collected in this trial with qualified researchers to help facilitate product development or enhancements in research that is not directly related to the study objectives. The informed consent explains this to the study subject.

# 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the study sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits

- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The principal investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number, and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

# 13.4 Sponsor and Monitoring Responsibilities

The study sponsor will select principal investigators that are qualified by education, training, and experience to assume responsibility for the proper conduct of this clinical trial.

The study sponsor is financially funding this clinical trial and will compensate the investigator and/or the institution(s) at which the study is conducted in accordance with a signed clinical trial agreement.

The study sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and wellbeing of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study

is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate study sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written, and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

## 13.5 Regulatory Documentation and Records Retention

The investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the study sponsor and the investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.

Additionally, the investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the study sponsor. If the investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the study sponsor must be notified, and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

# 13.6 Quality Assurance and Quality Control

The study sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the study sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the study sponsor with the investigator/institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

• Investigations are conducted in compliance with Good Clinical Practices; international and national regulations, laws and guidelines; the conditions of approval imposed by reviewing IRBs/IECs or regulatory authorities; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki The SOPs of the study sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations shall apply.

 Notifications and timelines for reporting protocol deviations should be based upon applicable ethics committee requirements.

The investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. The investigator is not allowed to deviate from the protocol except to protect the rights, safety, and wellbeing of human subjects under emergency circumstances. Emergency deviations may proceed without prior approval of the sponsor and the IRB/IEC, but shall be documented and reported to the sponsor and the IRB/IEC as soon as possible. Deviations from this protocol, regulatory requirements, and/or GCP must be recorded and reported to the sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Failure to implement identified corrective and preventative actions may result in site closure by the sponsor. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC. The investigator must provide documentation of the IRB/IEC approval to the study sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the package insert, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. Any additional requirements imposed by the EC or regulatory authority shall be followed. At the end of the study, the investigator must notify the IRB/IEC about the study's completion. The IRB/IEC also must be notified if the study is terminated prematurely. Finally, the investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject. The obtaining of consent shall be documented before any procedure specific to the clinical investigation is applied to the subject.

The investigator must have a defined process for obtaining the required consent. Specifically, the investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the investigator, and if required by local regulation, other qualified personnel. The investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and sponsor-designated personnel. The investigator must keep the original, signed copy of the consent (file in subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

The study sponsor assures that the key designs of this protocol will be registered on public databases where required by current regulations, and, as applicable, results will be posted.

#### 15 REFERENCES

## 15.1 Regulations and Standards

The following references may be applicable in whole or in part for this clinical trial.

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products -Guidance for clinical investigations
- EN ISO 14155:2020 Clinical Investigation of Medical Devices for Human Subjects -Good Clinical Practice
- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards

- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators

### 15.2 Scientific and Other References

Truong TN, Graham AD, Lin MC. Factors in Contact Lens Symptoms. Optometry and Vision Science. 2014; 91 (2): 133-141. doi: 10.1097/OPX.000000000000138









